CLINICAL TRIAL: NCT06872320
Title: The Influence of Probiotics on Metabolome and Heart Rate Variability in Heart Failure of Structure Heart Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202301449A3
Record Dates: First submitted 2024-11-28; First posted 2025-03-12 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-09

CONDITIONS: Congenital Heart Disease; Dysbiosis; Malnutrition, Child; Probiotics; Metabolome
MeSH Terms: conditions — Heart Defects, Congenital; Dysbiosis; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: One arm: participants will be stratified into two stratum and then assigned to one of the following double-blind treatment in a ratio of 2:1 at the randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Second arm:
  1. Serum NT-proBNP level: more than 25% decline of the level at entrySerum NT-proBNP level: more than 25% decline of the level at entry.
  2. The size of cardiac chambers, cardiac function, and shunt by echocardiography;
  3. Circulating levels of proinflammatory cytokines- TNF-α, IL-6, and IL-10 by multiplex immunoassay;
  4. Metabolomics study for heart failure patients with and without end-point improvement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus Rhamnosus (Active Comparator): Lactobacillus Rhamnosus (More than 1 billion colonies), Maltodextrin, Magnesium Stearate
  Interventions: Drug: Placebo
- placebo (Placebo Comparator): Maltodextrin, Magnesium Stearate
  Interventions: Drug: Lactobacillus Rhamnosus

INTERVENTIONS:
Drug: Lactobacillus Rhamnosus — Lactobacillus Rhamnosus (Lactobacillus Rhamnosus, MoProbi-LR Capsules, Drug permit license 052531); Age < 2 years old: 1/2 capsule once daily for 24 weeks per oral Age ≥ 2 years old: 1 capsule once daily for 24 weeks per oral
  Arms: placebo
Drug: Placebo — Maltodextrin comparable in color. Age < 2 years old: 1/2 capsule once daily for 24 weeks per oral Age ≥ 2 years old: 1 capsule once daily for 24 weeks per oral
  Arms: Lactobacillus Rhamnosus

SUMMARY:
Poor body weight gain and failure to thrive is a very common condition in patients with congenital heart disease (CHD) with advanced HF and/or cyanosis, which are considered a predictor of morbidity and complicate the prognosis of CHD. Studies have been carried out an attempt to discover the mechanisms to improve the therapies and the prognosis of these patients. Some of these studies give the hypothesis that the gastrointestinal tract, more precisely the intestine, can collaborate with metabolome. Extra-intracardiac shunt and HF lead to hypoperfusion and cyanotic heart disease leads to hypoxia. These two conditions make the gastrointestinal tract of these patients to become more mal-absorption to food. Consequently, the poor intestinal microcirculation and resultant dysbiosis may contribute to poor body weight gain and the worsening of prognosis. As known, probiotics can help to maintain or recover the microbiota and maintain a healthy intestinal barrier. In view of the importance of microbiota to the metabolism and the possible beneficial effect in the prognosis of heart-failure patients and the performance of microbiota in maintenance of intestinal barrier, this study has as primary objective to verify the influence of supplementation of the probiotic Lactobacillus Rhamnosus in the patients with CHD.

Malabsorption and dysbiosis in patients with CHD Poor body weight gain and failure to thrive is a very common condition in patients with congenital heart disease (CHD). Dysbiosis occurs in patients with CHD. Such dysbiosis and intestinal barrier dysfunction may become worsen after they underwent cardiopulmonary bypass, and complicate the prognosis of CHD.

Probiotics and Metabolome in Heart failure Cumulative evidence shows increasing importance of microbiota and cardiovascular disease and health. Metabolomic changes are found in CHD patients with hypoxia. It is suggested that Lactobacillus strains function to promote cardiovascular-related conditions. However, the effect of probiotic administration on CHD remains controversial. The investigators propose that hypothesis that Lactobacillus Rhamnosus directly improve the body weight gain and indirectly improve the outcome of patients with CHD. Accordingly, the investigators initiate this clinical trial to testify the beneficial effect of Lactobacillus Rhamnosus on CHD.

DETAILED DESCRIPTION:
Overall Design The present study will be a clinical trial compounded by two parallel arms, randomized, double-blind (researcher-patient), placebo-controlled, in patients with HF (HF) of varying degrees of functional class according the New York Heart Association (NYHA) or ROSS. There will be 120 subjects recruited, including two stratums (Strata 1, n= 90 and Strata 2, n= 30). Eighty of them (Strata 1 n= 60, Strata 2 n= 20) will receive probiotics, and forty (Strata 1 n= 30, Strata 2 n= 10) will receive placebo. These patients will be accompanied during 24 weeks and should take one capsule every day during the study. In the beginning and middle of the study and at the end, venous blood sample will be collected of each patient for laboratory measurement of TNF-α, interleukin (IL)-1, 6, and 10, NT-pro-B-type natriuretic peptide (BNP), and C-reactive protein (CRP). An anthropometric evaluation will be performed with measurements of weigh, height, arm circumference, triceps skin fold. According to nutritional status, it will be calculated the caloric and protein needs of each patient and, to monitor the consumption, in each consult will be applied the 24-hour food recall and calculated the consumption from it. In order to measure the appetite of the patients, in each consult, an appetite questionnaire will be applied. Before randomization, enrolled subjects will be categorized based on their HF severity secondary to volume/pressure overload, medications, and pulse oximeter for cyanotic heart disease.

1. Study type: interventional
2. Condition or disease: congenital heart disease, including structure, valvular heart disease and cardiomyopathy, with ejection fraction≥ 35%)
3. Intervention/treatment: dietary supplement with probiotics; others with placebo
4. Phase: not applicable
5. Estimated enrollment: 150 participants
6. Allocation: stratified randomization, according to NYHA/ROSS HF classification
7. Intervention model: parallel assignment
8. Masking: double (participant, investigator)
9. Primary purpose: treatment for 24 weeks
10. Final study follow-up: 3 months
11. Official title: Effect of Lactobacillus Rhamnosus in Patients with Congenital Heart Disease- randomized, double-blind study
12. Study start date: Jan 1, 2024
13. Estimated primary completion date: Dec 31, 2026
14. Estimated study completion date: Jan 30, 2025 (follow-up)
15. Study location: single center at Kaohsiung Chang Gung Memorial Hospital, Taiwan

Aim 1: To characterize the HRV pattern and metabolome in small children with CHD based on the severity of HF (1st year).

i. To recruit participants who meet the study criteria and substrate them into mild and severe CHD-HF.

ii. To study echocardiography to evaluate the cardiac function at indicated time points.

iii. To obtain plasma samples for HF markers. iv. To perform HRV study on patients and to characterize the HRV pattern based on HF severity.

Aim 2: To explore the metabolome and to elucidate the relationships between metabolome and HRV in CHD-HF (2nd year).

i. To investigate metabolome in the study population. ii. To characterize the "bad" and "good" metabolome according to the changes of HRV and/or CHD-HF severity.

iii. To examine the relationships between metabolome and HRV.

Through aims 1 and 2 prescribed above, the investigators will be able to understand metabolome and HRV status in CHD with various HF.

Aim 3: To explore the changes of CHD-HF, HRV, and metabolome after probiotics Lactobacillus Rhamnosus. This clinical trial protocol was reviewed and approved by the Taiwan Food and Drug Administration (MoProbi-LR Capsules, Drug permit license 052531 ) usage (3rd year).

i. To explore the changes of clinical parameters in CHD-HF after probiotics usage.

ii. To analyze the alteration in HRV pattern before and after probiotics iii. To analyze the alteration in metabolomic profile before and after probiotics.

iv. To examine the beneficial role of probiotics in CHD-HF.

Treatments

1. Study populations Inclusion/Exclusion and Withdraw Criteria： Inclusion

   Criteria:

   1-1. Patients at ages ≤ 3 years old with congenital structure/valvular heart disease and cardiomyopathy with varying degrees of HF NYHA/ROSS functional class and ejection fraction ≥ 35% by echocardiography at the entry of study; 1-2. No recent 1-month hospitalizations for HF decompensated; 1-3. Have signed the Free and Informed Consent Form Exclusion Criteria: 1-3-1. CHD with NYHA functional class IV or ejection fraction 35%; 1-3-2. Do not accept to participate in the study or do not sign the Free and Informed Consent Form; 1-3-3. Have used antibiotics and/or corticosteroids and/or other formula containing probiotics in the last 30 days prior enrollment; 1-3-4. Clinical conditions that can affect the inflammatory profile such as inflammatory bowel disease, arthrosis, among others; 1-3-5. Chronic severe diarrhea (> 2 weeks; > 5 times/day) in the last 3 months; 1-3-6. Have been submitted to a cardiac surgery or other surgery in the last 3 months; 1-3-7. Severe lactose intolerance; 1-3-8. Profound anemia (WBC>15000, Hb< 8 ) or hematologic disorder, severe hepatic dysfunction (GPT>100), renal function (Cr>1.5), abnormal stool analysis or active infection status (CRP> 10).
2. Withdrawal criteria:

   The anticipated circumstances under which the Principal Investigator (PI) may terminate a participant's participation in the study, regardless of the participant consent; 2-1. Poor cooperation in treatment or assessment 2-2. Take other probiotics for more than 2 months 2-3. Receive major cardiovascular surgery during the treatment period 2-4. Severe infection occurs and lasts for more than 1 month during the treatment period 2-5. Severe adverse effects after taking probiotics (after other possible cause being ruled out) such as severe diarrhea or allergy/skin rash If the condition mentioned above occurs 3 months after entry of the trial study, the data of the participant will be recorded and finally analyzed. If the condition occurs less than 3 months since the entry, the participant will be dropped out from this trial after tremendous evaluation. If so, the related information, data, and assessment will be completely deleted. The consequences of a participant's decision to withdraw from non-exempt research and the procedures for orderly and safe termination of her/his/their participation.

   Any condition that the participant or the guarder unwilling to stay in the study.
3. Treatment Administration Oral intake once daily : Lactobacillus Rhamnosus (Lactobacillus Rhamnosus, MoProbi-LR Capsules, Drug permit license 052531 ); other: placebo Age ≦ 2 years old: 1/2 capsule once daily for 24 weeks per oral Age ≥ 2 years old: 1 capsule once daily for 24 weeks per oral Allowance: total discontinued treatment less than 30 days, or successive discontinuation less than 14 days.

   3-1 Treatment arms One arm: participants will be stratified into two stratum and then assigned to one of the following double-blind treatment in a ratio of 2:1 at the randomization.

   3-2 Treatment assignment and randomization All participants will be stratified into two stratum by HF NYHA/modified ROSS10 functional class and pulse oximeter to ensure a balanced distribution of heart disease severity. Strata 1: HF NYHA/ROSS functional class I and/or pulse oximeter≥ 90%; Strata 2: HF NYHA/ROSS functional class II-III and/or pulse oximeter≧90%. PI will confirm that the participant fulfills all the inclusion/exclusion criteria and then assigns a randomization number to the participant, which will be used to link the participant to the treatment and will specify a unique medication number. The randomization numbers will be generated to ensure that treatment assignment is unbiased and concealed from participants and Investigator staff. A participant randomization list will be produced by the IRT/or the statistic center of KCGMH using a validated system that automates the random assignment of patient numbers to randomization numbers. The randomization scheme for participants will be reviewed and approved by IRB and the statistic center 3-3. Treatment blinding

   This trial is a randomized, double-blind, active controlled study. Participants, Investigator, staff, persons performing the assessment and data analysts will remain blind to the identity of the treatment from the time of randomization until database lock using the following methods:

   3-3-1.Randomization data will be kept strictly confidential until the time of unblinding, and will not be accessible by anyone involved in the study with the following exceptions: A. The independent and unblinded satisfaction, programmer and data personnel who are involved in preparing safety and efficacy interim analysis report for the DMC. These personnel will not be involved in any other trial conduct related activities.

   B. The DMC members A double-dummy design is used because the identity of the investigational treatment cannot be disguised, as the drug products are visibly different.

   The identity of the treatments will be concealed by the use of investigational treatment that are all identical in packaging, schedule of administration, appearance, taste and odor.

   Unblinding will only occur in the case of patient emergencies, at the time of the interim analysis, and at the conclusion of the study.

   3-3-2. Concomitant Therapy：Some patients may take anti-congestive medication (e.g., captopril, Lasix, digoxin) or anti-platelet (e.g., aspirin) or anti-coagulation (e.g., coumadin) prescribed to control underlying cardiovascular status.
4. Efficacy Assessments 4-1. Primary end-point：Body weight percentile (BWP) gain: increase of BWP from the base line to the end of 24-wk treatment (increase in 15th percentile for those patients with prior BWP more than 10th percentile or Strata 1, and 10th percentile for those with prior BWP ≤10th percentile or Strata 2); the measurement of BW percentile according to the Taiwan children growth reference.

   4-2. Secondary end-point 4-2-1. Decrease of cardiac chamber enlargement: The body surface area-normalizing size of cardiac chambers as well as cardiac function, and shunt by echocardiography or 4-2-2. Serum NT-proBNP level: more than 25% decline of the level at entry. 4-3. Surrogate markers 4-3-1. Circulating levels of proinflammatory cytokines- TNF-α, IL-6, and IL-10 by multiplex immunoassay.

   4-3-2. Metabolomics study for HF patients with and without end-point improvement (for future study if inadequate funding budget).

   4-3-3. All these assessments will be measured and recorded at indicated time points as listed in time-event scheme, and will be statistically analyzed at the end of this study
5. Schedule of Activities From being screened to the end of the study, every participant must visit clinics 9 times for vital sign check, physical examination, and body weight and height measurements. Echocardiography and 12-lead EKG as well the investigators nutrition consultation and intervention will be performed at screening stage, at 1 and 3 months after entry the study, and at the end of the treatment. Blood test and stool sampling will be done 3 times at screening and at the middle and end of treatment. Stool analysis will be executed at screening and at the safety follow-up visit.
6. Safety Assessments 6-1. Blood tests including hemogram (CBC/DC), ALT, AST, Cr, sodium, potassium, chloride, CRP, vein blood gas, blood culture and stool culture.

   6-2. Stool analysis and stool culture at the beginning and the end of study. 6-3. Serious adverse effect such as severe allergy or diarrhea. 6-4. All these assessments will be performed and recorded at indicated time points before the entry or at the beginning, middle, and the end of study. The participant will be allowed to participate if there is no stool occult blood, leukocyte, or pus and negative stool culture.
7. Adverse event reporting

   Dr Lin will report SAEs to the IRB of Chang Gung Medical Foundation according to the Serious Adverse Event Reporting Procedures and Guidelines as posted in the Clinical Trials Resource on the website of Chang Gung Medical Foundation IRB. SAE reports to the IRB should include the following information when calling the Medical Monitor:

   7-1. Date and time of the SAE 7-2. Date and time of the SAE report Name of reporter 7-3. Call back phone number Affiliation/Institution conducting the study Protocol number.

   7-4. Title of protocol 7-5. Description of the SAE, including attribution to drug and expectedness
8. Materials and Methods 8-1. Measurement of Echocardiography and Cardiac Output Echocardiography will be performed for all offspring without any harm after care sedation and removal of chest hair. Any follow-up parameters will be also collected. Echo machine Philips IE33 and EPIQ with transducer S5, S8 or S12 will be used to evaluate all recruited subjects to measure cardiovascular function and cardiac output. Meanwhile, clinical hemodynamic parameters such as SBP, DBP and MBP and arterial blood gas data if any will be collected. Echo machine will be used to evaluate all recruited subjects to measure each cardiovascular segment as well 2D Simpson's method, tissue doppler imaging and global longitudinal strain.

8-2. Metabolic Profile (Alternative method to assess vascular function) Serum/plasma vascular profile, including vascular endothelial growth factor (VEGF)-A, soluble vascular cell adhesion molecule (sVCAM), soluble intercellular adhesion molecule (sICAM), E-selectin, P-selectin, endothelin-1, thromboxane A2 (TXA2), monocyte chemoattractant protein (MCP)-1, TNF-α, and interleukin (IL)-1β will be served as an alternative index for vascular injury (as a surrogate evidence of endothelial dysfunction) and indicates possible vascular injury and/or undergoing vascular repair. Meanwhile, plasma and urine samples from recruited human subjects will be simultaneously assayed for the levels of asymmetric dimethylarginine (ADMA) and nitric oxide (NO) as another surrogated index of vascular injury/endothelial activation/endothelial dysfunction by ELISA kit.

8-3. HF markers

HF markers include serum NT-proBNP level, and sodium. Meanwhile, osmolality, renal function will be also checked. and will be used as secondary endpoints:

Surrogate markers 8-3-1. Circulating levels of proinflammatory cytokines- TNF-α, IL-6, and IL-10 by multiplex immunoassay.

8-3-2. Metabolomics study for HF patients with and without end-point improvement (for future study if inadequate funding budget).

8-4. HRV Heart rate variability (HRV) is used as an indirect autonomic assessment provides prognostic information when measured over short time periods in patients with heart failure. VLF power is an independent risk predictor in patients with CHF.11 SDAAM declines as patient status decompensate. Continuous long-term SDAAM may be a useful tool in the clinical management of patients with chronic heart failure.12 In the Multi-Ethnic Study of Atherosclerosis (MESA),13 a population-based study of subclinical cardiovascular disease in adults aged 45 to 84 years, the investigators measured the heart rate variability using a standard 30-second, 12-lead electrocardiogram to measure the SDNN and the root mean square of successive differences in RR intervals (RMSSD). In pediatric CHD, tachycardia with readily diaphoresis are frequently observed in CHD patients with severe HF. Thus, the investigators would like to assess the HRV in such population and will used it as the HF index.

8-5. Metabolome Profile Metabolome profiles will be focus on long-chain and short-chain fatty acids (LCFAs and sCFAs) and TMAO as well as HOMA-IR index (Homeostasis model assessment-insulin resistanc index (central lab code: L72-314 and L72-496), HbA1c, fasting sugar, and DM lipid profile (tota cholesterol, triglycerides and cholesterol subtypes). The plasma will be collected and stored at -80℃. Gas chromatography mass spectrometry (Agilent 7890B) with an automated sample will bused to measure plasma FA concentrations. A DB-FFAP column (30 m × 0.25 mm, 0.25 µm Agilent Technologies) will be used for chromatographic separation. The injection volume will be 1 µL in a split ratio of 5:1 at 240°C. Helium will be the carrier gas with a flow rate of 1 mL/mi through the column; the front inlet purge flow was 3 mL/min. An internal standard will b 2-ethylbutiric acid. The GC mass spectrometry will be operated using an ionization voltage of 7 eV with an ion source temperature of 230℃. Six SCFAs including acetate, propionate, isobutyrate butyrate, isovalerate and valerate in the gas-phase ions will be detected 8-6. Compositional of Gut Microbiota analysis DNA will be extracted from the gut microbiome of frozen fecal samples with QIAamp DNA Stool Mini Kit (Qiagen) according to the manufacturer's protocol. DNA will be quantified by a NanoDrop ND-1000 Spectrophotometer. The variable regions 3-4 (V3-4) of small subunit rRNA (16S rRNA) gene will be amplified with primers 341F (50 - CCTACGGGNGGCWGCAG-30 ) and 805R (50 -GACTACHVGGGTATCTAATCC-30 ). The PCR reactions will be carried out in reactions with PCR Master Mix, primers and template DNA. Thermocycler will be used the following protocol. Amplicons will be analyzed and sequenced using the illumine MiSeq paired-end sequencing platform. 97% sequences similarity will be clustered to the same operational taxonomic units (OTUs) by Uparse software. Taxonomic annotation of the OUT representative sequences will be performed using the Ribosomal Database Project (RDP) classifier retrained on the Greengenes 16S rRNA gene database. The level of alpha and beta diversity in the samples will be analysis by QIIME software.

8-7. Real Time RT-PCR for specific gene confirmation Transcripts of 1μg total RNA from specimens will be reverse-transcribed and the resultant cDNA will be amplified by ABI 7500 Sequence Detector for real-time reverse transcriptase- polymerase chain reaction for target genes selected from the result of transcriptome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at ages ≤ 3 years old with congenital structure/valvular heart disease and cardiomyopathy with varying degrees of HF NYHA/ROSS functional class and ejection fraction ≥ 35% by echocardiography at the entry of study;
2. No recent 1-month hospitalizations for HF decompensated;
3. Have signed the Free and Informed Consent Form.

Exclusion Criteria:

1. CHD with NYHA functional class IV or ejection fraction < 35%;
2. Do not accept to participate in the study or do not sign the Free and Informed Consent Form;
3. Have used antibiotics and/or corticosteroids and/or other formula containing probiotics in the last 30 days prior enrollment;
4. Clinical conditions that can affect the inflammatory profile such as inflammatory bowel disease, arthrosis, among others;
5. Chronic severe diarrhea (> 2 weeks; > 5 times/day) in the last 3 months;
6. Have been submitted to a cardiac surgery or other surgery in the last 3 months;
7. Severe lactose intolerance;
8. Profound anemia (WBC> 15000, Hb< 8 ) or hematologic disorder, severe hepatic dysfunction (GPT> 100), renal function (Cr> 1.5), abnormal stool analysis or active infection status (CRP> 10).

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentile of body weight gain | From enrollment to the end of treatment an average of 24 weeks.
  The difference of body weight percentile from the enrollment as the base line to the end of 24-wk treatment (Body weight percentile will be calculated according to the Taiwan children growth reference：https://growth.healthinfo.tw )

SECONDARY OUTCOMES:
Decrease of cardiac chamber enlargement. | The difference of following measurements from the enrollment as the base line to the end of 24-wk treatment
  The z scores of cardiac chambers (i.e., left and right ventricles and atria) using body surface area-normalization
The cardiac function | The difference of following measurements from the enrollment as the base line to the end of 24-wk treatment
  The cardiac function: ejection fraction (%), global longitudinal strain (%) of left ventricle, LA strain (%), or the ratio of mitral e/e', and Qp/Qs shunt by echocardiography
Serum NT-proBNP leve | The difference of following measurements from the enrollment as the base line to the end of 24-wk treatment
  Serum NT-proBNP level

OTHER OUTCOMES:
Circulating levels of proinflammatory cytokines | The difference of following measurements from the enrollment as the base line to the end of 24-wk treatment
  Circulating levels of proinflammatory cytokines- tumor necrosis factor-α (pg/ml), interleukin-6 (pg/ml), and interleukin-10 (pg/ml) by multiplex immunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital and Chang Gung University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP